CLINICAL TRIAL: NCT04086693
Title: Peripheral Intravenous Catheter Securement With Tissue Adhesive Compared to Conventional Dressing: A Randomized Controlled Trial
Brief Title: Peripheral Intravenous Catheter Securement With Tissue Adhesive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Amit Bahl, Director Emergency Medicine Ultrasound, Corewell Health East
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-188
Record Dates: First submitted 2019-09-09; First posted 2019-09-12 (Actual); Results first posted 2021-02-01 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Vascular Access Devices
Keywords: intravenous access; vascular access; IV survival; IV catheter complication

STUDY DESIGN:
Intervention Model Description: Randomized controlled, parallel assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard IV dressing (Active Comparator): Polyurethane dressing with clear tape
  Interventions: Device: Standard IV dressing
- Standard IV dressing plus Adhezion SecurePortIV (Experimental): Polyurethane dressing with clear tape plus Adhezion Biomedical SecurePortIV (a tissue adhesive peripheral IV securement device).
  Interventions: Device: Standard IV dressing plus a tissue adhesive peripheral IV securement device

INTERVENTIONS:
Device: Standard IV dressing — Polyurethane and clear tape dressing used to secure peripheral IV
  Arms: Standard IV dressing
Device: Standard IV dressing plus a tissue adhesive peripheral IV securement device — Polyurethane dressing with clear tape plus a tissue adhesive peripheral IV securement device used to secure peripheral IV
  Other Names: Adhezion SecurePortIV
  Arms: Standard IV dressing plus Adhezion SecurePortIV

SUMMARY:
This clinical trial will compare survival of peripheral intravenous (IV) catheters for patients with a standard IV site dressing alone to patients with standard IV dressing plus Adhezion Biomedical SecurePortIV Catheter Securement Adhesive. Emergency room patients who already have IVs may be considered for inclusion. Eligible patients will be approached and, if they are interested in participating, their informed consent will be obtained. Participation will continue for up to 7 days. During this time, the patient will experience:

* Assessment of their currently placed peripheral IV catheter, to assess if it is functioning
* Assignment to one of two study groups (standard IV dressing or standard IV dressing plus Adhezion Biomedical SecurePortIV Catheter Securement Adhesive). This is called randomization and group assignment is by chance, like the flip of a coin
* Daily assessment of the IV catheter and site for complications (such as infection or phlebitis), removal, and medications being administered.

DETAILED DESCRIPTION:
Patients admitted from the Emergency Department (ED) to a progressive floor, or patients admitted from ED to any floor type with express approval from the Principal Investigator are eligible participants. Research staff will approach patients admitted to the progressive floors (or other floors when identified by PI) based on screening of the electronic medical record. These patients are approached by research staff when physically in the emergency department waiting for a room assignment. If the patient agrees to participate in the trial, the study subject will approached for consent by the research staff. Research staff will confirm functionality of the existing peripheral IV previously placed by ED staff. The assessment will include observing for blood return into the tubing upon aspiration and/or unobstructed flush with a minimum of 1-2 ml of normal saline. Staff will also observe the site for any signs of redness or tenderness. A tourniquet may be applied as needed. If the patient is actively receiving an infusion, the drip will briefly be halted to evaluate for functionality. Functionality will be assessed with the existing dressing in place. If the catheter is functional and free of any signs of complications, study subjects will be randomized by a computer generated 1:1 envelope system to either the control group: polyurethane dressing + clear tape or the experimental group: polyurethane dressing + clear tape + tissue adhesive. The tissue adhesive is not standard of care at Beaumont. For the control group, the polyurethane dressing will be gently removed. Dressing will be removed carefully to minimize any potential dislodgments or skin injury. The site will be evaluated for oozing or blood and as needed cleaned with sterile gauze. Once the site is completely dry, a new polyurethane dressing will be applied and reinforced with tape in a standard fashion. Once securement is complete, functionality will be reassessed per protocol above. For the experimental group, the existing securement will be gently removed. There are not special steps required for removing the dressing with the tissue adhesive. The IV catheter is secured and the dressing is removed gently. The site will be evaluated for oozing or blood and as needed cleaned with sterile gauze. Once the site is completely dry, the tissue adhesive will be applied. A new standard polyurethane dressing will be applied and tape will be applied per the standard approach. Once securement is complete, functionality will be reassessed. The time of the new dressing application will be noted as time zero. Catheter dwell time will begin at this point. Additional data variables collected at the initial assessment include: demographics such as age, sex, international normalized ratio (INR) >1.5, platelets < 50, insertion site details, hours from insertion to recruitment, inserter credentials.

Follow-up Assessment:

After initial assessment, the catheter will be assessed by the research team every 24 hours as long as the patient is hospitalized up to 7 days or 168 hours. At each follow up interval the researcher notes the date /time of evaluation and assesses for any signs and symptoms of complications and functionality of the device. A catheter is functional if the IV flushes without resistance. Complications include infiltration, phlebitis, dislodgement, oozing fluid/blood, purulent drainage, or occlusion. Catheters will be assessed daily for signs and symptoms of complications. Any signs or symptoms of complications or lack of functionality will be reported to the patient's primary care team so that management of the IV catheter can be addressed. If the catheter was identified to have any signs or symptoms of complications during follow-up assessment the date and time of observation of the complication will be documented in the data collection tool and the primary team will be notified of the complication. If the catheter was removed prior to the follow-up assessment then the IV removal time and the reason for removal will be obtained through chart review. For all catheters removed due to a complication, re-insertion attempt data will be tracked through the medical record in the nursing section for venous lines and need for reinsertion of the IV or escalation to a midline, peripherally inserted central catheter (PICC), or central venous catheter (CVC) will be noted. If the patient is discharged prior to the time of follow-up assessment then the time of discharge will be documented and the IV will be presumed functional until time of discharge unless otherwise noted in the chart.

The medication administration record will be queried for all medications given through each catheter with specific attention to antibiotics and anticoagulants. Vesicants/irritants that are generally given via central line or considered caustic to the vessel will be noted in both groups. Number of doses will be recorded. Additional data gathered by research staff on follow-up evaluation includes: dwell time in days/hours, hospital length of stay, and number of peripheral IVs for duration of stay.

ELIGIBILITY:
Inclusion Criteria:

1. Greater or equal to 18 years of age
2. Admission from the Emergency Department (ED) to a progressive floor, or Admission from ED to any floor type with express approval from the Principal Investigator
3. IV placement in the antecubital fossa, forearm, wrist or hand
4. IV placement in the ED
5. Enrollment within 8 hours of IV insertion
6. 18 or 20 gauge 1.16 inch IV catheter
7. Expected hospital admission >48 hours

Exclusion Criteria:

1. Patients with ultrasound-guided IV insertions
2. Alternate site of cannulation
3. Voluntary withdrawal
4. Patients with a non-standard polyurethane dressing
5. Known allergy to cyanoacrylate or formaldehyde

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2020-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Bahl, MD, Principal Investigator — Corewell Health East
Locations (1):
- Beaumont Health System, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 350
Period: Overall Study
Arm/Group | Standard IV Dressing | Standard IV Dressing Plus Adhezion SecurePortIV
Started | 175 | 175
Completed | 174 | 171
Not Completed | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard IV Dressing | Standard IV Dressing Plus Adhezion SecurePortIV | Total
Number analyzed (Participants) | 174 | 171 | 345
Age, Continuous [Median (Standard Deviation); unit: years] | 68.0 (15.3) | 68.8 (15.4) | 68.4 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 73 | 152
  Male | 95 | 98 | 193
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: IV Catheter Survival
Description: Number of participants with all-cause functional failure of the catheter. Failure is defined by loss of patency (resistance to flush with minimum 1-2 ml normal saline, or lack of blood return to tubing on aspiration) or presence of complications requiring removal (any level of pain or tenderness, changes in skin color (blanching or erythema), changes in skin temperature (hot or cold), edema, induration, leakage of fluid or purulent discharge from the puncture site, or other dysfunction). Function is assessed daily by research staff.
Time Frame: 7 days or discharge, whichever occurs sooner
Measure: Count of Participants; unit: Participants
Arm/Group | Standard IV Dressing | Standard IV Dressing Plus Adhezion SecurePortIV
Number analyzed (Participants) | 174 | 171
Participants | 66 | 55

2. Secondary Outcome: Mean Catheter Survival Duration
Description: Mean catheter survival duration in days
Time Frame: 7 days or until discharge, whichever occurs sooner
Population: Numbers of participants reflect those fulfilling 48 hour dwell per protocol
Measure: Mean (Full Range); unit: days
Arm/Group | Standard IV Dressing | Standard IV Dressing Plus Adhezion SecurePortIV
Number analyzed (Participants) | 141 | 142
days | 5.43 [0 to 7] | 5.97 [0 to 6.71]

3. Secondary Outcome: Cause-specific IV Failure
Description: Number of participants with IV catheter failures by specific cause, including infiltration, phlebitis, dislodgment, leaking, infection, and occlusion. IV failure is assessed daily by research staff and by chart review, post patient discharge
Time Frame: 7 days or until discharge, whichever occurs sooner
Measure: Count of Participants; unit: Participants
Arm/Group | Standard IV Dressing | Standard IV Dressing Plus Adhezion SecurePortIV
Number analyzed (Participants) | 174 | 171
Participants
  Infiltration | 23 | 26
  Phlebitis | 13 | 10
  Dislodgement | 8 | 3
  Leaking | 31 | 24
  Occlusion | 1 | 3
  Death of Participant | 1 | 1
  Other | 1 | 1
  Completion of Therapy | 96 | 103

ADVERSE EVENTS:
Time Frame: Adverse event data was collected on each patient from IV insertion until IV removal for a maximum of 7 days.
Arm/Group | Standard IV Dressing | Standard IV Dressing Plus Adhezion SecurePortIV
All-Cause Mortality (participants affected / at risk) | 1/174 | 1/171
Serious Adverse Events (participants affected / at risk) | 0/174 | 0/171
Other Adverse Events (participants affected / at risk) | 0/174 | 0/171

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-16): https://cdn.clinicaltrials.gov/large-docs/93/NCT04086693/Prot_SAP_001.pdf